CLINICAL TRIAL: NCT06245395
Title: Virtual Reality as Distraction Analgesia and Anxiolysis for Pediatric Otolaryngology Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WalterReedNMMC - ENT
Record Dates: First submitted 2024-01-29; First posted 2024-02-07 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Virtual Reality; Otolaryngology

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Arm (Active Comparator): Pediatric patient receiving Virtual Reality during the otologic procedure.
  Interventions: Device: Virtual Reality
- Standard of Care Arm (No Intervention)

INTERVENTIONS:
Device: Virtual Reality — Meta Quest 2 Headset
  Arms: Virtual Reality Arm

SUMMARY:
The primary aim of this randomized controlled trial is to determine the efficacy of Virtual Reality in pediatric otolaryngology clinics as distraction analgesia and anxiolysis for patients undergoing otologic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients, ages 7-17 years old, undergoing an in-office microscope ear examination with possible debridement/instrumentation by a single fellowship trained neurotologist .

Exclusion Criteria:

* 1) patients with a history of chronic pain disorders 2) developmental delay including autism spectrum disorders 3) neurologic or seizure disorders 4) visual impairment 5) claustrophobia

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Wong-Baker FACES Pain Scale | during the in clinic procedure
Subjective Units of Distress Scale | during the in clinic procedure

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Tolisano, MD, Principal Investigator — WRNMMC
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided